CLINICAL TRIAL: NCT04310592
Title: A Phase I Multi-dose Study of Human Placental Hematopoietic Stem Cell Derived Natural Killer Cells (CYNK-001) with or Without Recombinant Human Interleukin-2 (rhIL-2) in Adults with Primary or Secondary Acute Myeloid Leukemia (AML) in Morphologic Complete Remission with Minimal Residual Disease (MRD) or Relapsed/refractory (R/R) AML
Brief Title: Natural Killer Cell (CYNK-001) Infusions in Adults with AML
Acronym: CYNK001AML01
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business reasons
Sponsor: Celularity Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CYNK-001-AML-001
Record Dates: First submitted 2020-03-12; First posted 2020-03-17 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2023-03

CONDITIONS: Leukemia; Leukemia, Myeloid; Leukemia, Myeloid, Acute; Neoplasms by Histologic Type; Neoplasms; Immunosuppressive Agents; Immunologic Factors; Physiological Effects of Drugs; Alkylating Agents; Antimetabolites, Antineoplastic; Antiviral Agents; Analgesics, Non-narcotic; Anti-infective Agents; Analgesics; Peripheral Nervous System Agents; Hematologic Diseases; Hematologic Neoplasms; Leukemia in Remission; Relapsed Adult AML; Refractory AML
Keywords: CYNK-001; Acute Myeloid Leukemia; Acute Myelogenous Leukemia; allogeneic; allogeneic stem cell transplant; AML; cell therapy; cyclophosphamide; fludarabine; minimal residual disease; MRD; newly diagnosed AML; newly diagnosed acute myeloid leukemia; NK cells; natural killer cells; fludarabine phosphate; antineoplastic agents, alkylating; molecular mechanisms of pharmacological action; relapsed AML; refractory AML
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid; Leukemia, Myeloid, Acute; Neoplasms by Histologic Type; Neoplasms; Hematologic Diseases; Hematologic Neoplasms; Neoplasm, Residual

STUDY DESIGN:
Intervention Model Description: Experimental: Minimal Residual Disease (MRD) positive AML patients; Cyclophosphamide + Fludarabine + CYNK-001. On Days 0, 7, and 14, (and 21 in certain arms) CYNK-001 at 3 varying dose levels.
  Experimental: Relapsed/Refractory AML patients; Cyclophosphamide + Fludarabine + CYNK-001. On Days 0, 7, and 14, (and 21 at certain dose levels) CYNK-001 at 3 varying dose levels.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dose escalation/MTD or MPD determination in MRD positive AML patients (Experimental): Cyclophosphamide + Fludarabine prior to CYNK-001 on Days 0, 7, and 14; CYNK-001 at 3 varying dose levels.
  Interventions: Biological: CYNK-001
- Dose escalation/MTD or MPD determination in Relapsed/Refractory AML patients (Experimental): Cyclophosphamide + Fludarabine prior to CYNK-001 on Days 0, 7, and 14; CYNK-001 at 3 varying dose levels.
  Interventions: Biological: CYNK-001

INTERVENTIONS:
Biological: CYNK-001 — CYNK-001 is an allogeneic off the shelf cell therapy enriched for CD56+/CD3- NK cells expanded from human placental CD34+ cells.

SUMMARY:
This study will find the maximum tolerated dose or the maximum planned dose of CYNK-001 which contains natural killer (NK) cells derived from human placental CD34+ cells and culture-expanded. CYNK-001 cells will be given after lymphodepleting chemotherapy. The safety of this treatment will be evaluated, and researchers want to learn if NK cells will help in treating acute myeloid leukemia.

ELIGIBILITY:
Treatment Eligibility Screening Patient Inclusion Criteria

Patients must satisfy the following criteria to be enrolled in the study:

* Patient has eligible disease status:

  * Primary or Secondary acute myeloid leukemia (AML) Patients in first of second Morphological Complete Remission (CR), Morphological Complete Remission with incomplete hematologic recovery (CRi), or Morphologic Leukemia-free State (MLFS) as defined by the European LeukemiaNet (ELN) recommendations for AML Response Criteria (Dohner, 2017).
  * R/R diagnosis based on confirmed diagnosis with local pathology report following any reinduction/ salvage therapy ELN guidelines.

    1. Relapsed AML are defined as having relapsed after achieving ≥ 1 CR, including relapse after allogeneic stem cell transplantation (≥ 2 months after transplant).
    2. Refractory AML, defined as not achieving CR, CRi, or MLFS after 2 or more cycles of induction therapy (primary refractory) or not achieving CR after treatment for relapsed AML.
    3. Secondary AML (MDS transformation): Secondary AML patients are eligible to participate if they have received a minimum of one prior line of treatment for AML.
    4. Treatment-related AML: Treatment-related AML patients are eligible to participate if they have received a minimum of one prior line of treatment for AML.
* Patient with prior central nervous system involvement by malignancy are eligible provided that it has been treated and cerebral spinal fluid is clear for at least 2 weeks prior to start of Lymphodepletion Regimen.
* (MRD positive population only): Patient is minimal residual disease (MRD) positive, as assessed on bone marrow aspirate (BMA) by Multiparameter Flow Cytometry (MFC) at time of Treatment Eligibility assessment.

For the purposes of this study, MRD positivity is defined as greater than or equal to 0.1% blasts detected by MFC on BMA by the Sponsor-selected Central MRD analysis laboratory, where assay sensitivity allows for a Lower Limit of Detection (LOD) of 1 x 10-4 (0.01%) or lower.

* Patient is ≥ 18 and ≤ 80 years of age at the time of signing the Study informed consent form (ICF).
* Patient understands and voluntarily signs the Study ICF prior to any study-related assessments/procedures are conducted.
* Patient is willing and able to adhere to the study schedule and other protocol requirements.
* Performance status of Eastern Cooperative Oncology Group (ECOG) ≤ 2.
* Ability to be off immunosuppressive drugs for at least 3 days prior to the CYNK-001 infusion. Steroids at the equivalent of no more than 7.5 mg prednisone per day are permissible.
* Female of childbearing potential (FCBP)* must not be pregnant and agree to not becoming pregnant for at least 28 days following the CYNK-001. FCBP must agree to use an adequate method of contraception during the treatment period.

  * FCBP is a female who: 1) has achieved menarche at some point, 2) has not undergone a hysterectomy or bilateral oophorectomy or 3) has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months).
* Male Patients must agree to use a condom during sexual contact for at least 28 days following the last infusion of CYNK-001, even if he has undergone a successful vasectomy.

Treatment Eligibility Screening Patient Exclusion Criteria

The presence of any of the following will exclude the Patient from enrollment:

* Patient has any significant medical condition, laboratory abnormality, or psychiatric illness that would prevent the Patient from participating in the study.
* Patient has any condition including the presence of laboratory abnormalities which places the Patient at unacceptable risk if he or she were to participate in the study.
* Patient has any condition that confounds the ability to interpret data from the study.
* Patient has bi-phenotypic acute leukemia.
* Patient has acute promyelocytic leukemia (APL).
* Patient has inadequate organ function as defined below at time of Treatment Eligibility Period:

  1. Patient has aspartate aminotransferase (AST), alanine aminotransferase (ALT), or alkaline phosphatase ≥ 2.5 x the upper limit of normal (ULN).
  2. Estimated glomerular filtration rate (eGFR) < 30 mL/min/1.73 m2 as calculated using the Modification of Diet in Renal Disease Study equation (Levey, 2006) or history of an abnormal eGFR < 60 and a decline of > 15 mL/min/1.73 m2 below normal in the past year.
  3. Patient has a bilirubin level > 2 mg/dL (unless Patient has known Gilbert's disease).
* Patient has had prior treatment with biologic antineoplastic agents less than 7 days before first CYNK-001 infusion and at least 5 half-lives. (Exception will be granted for monoclonal antibodies that are known to have long half-lives, in which case a minimum of 2 weeks from last dose will be required). For agents that have known AEs occurring beyond these specified days after administration, this period must be extended beyond the time during which acute AEs are known to occur. Treating physicians are encouraged to discuss cases with the Medical Monitor.
* Patient is pregnant or breastfeeding.
* Patient has new or progressive pulmonary infiltrates or pleural effusion large enough to be detected by chest x-ray or CT scan within 2 weeks of first CYNK-001 infusion.
* Patient has active autoimmune disease other than controlled connective tissue disorder or those who are not on active therapy.
* Patient has had a Bone Marrow transplant < 60 days prior to screening or plans to have a transplant within the 28 day period following the first CYNK-001 infusion.
* Patient has a history of malignancy other than AML or other underlying hematologic conditions such as myelodysplastic syndromes (MDS) or myeloproliferative neoplasms (MPN) unless the Patient has been free of disease for greater than 3 years prior to CYNK 001 infusion. Exceptions will include the following malignancies:

  1. Basal cell carcinoma of the skin
  2. Squamous cell carcinoma of the skin
  3. Carcinoma in situ of the cervix
  4. Carcinoma in situ of the breast
  5. Incidental biological finding of prostate cancer (TNM stage of T1a or T1b)
  6. Superficial bladder cancer
  7. For patients with therapy-related AML, the underlying malignancy which led to secondary AML must be stabilized (not progressing) and not under active treatment.
* Patient has a history of severe asthma and is presently on chronic medications or has a history of other symptomatic pulmonary disease.
* Patient has the following prior history of GVHD:

Acute GVHD: Subjects with prior history of acute GVHD where signs and/or symptoms did not completely resolve (no clinical signs/symptoms and not on more than 7.5 mg of predinsone per day Chronic GVHD: Subjects with prior history of chronic GVHD where signs and/or symptoms did not completely resolve (no clinical signs/symptoms and not on more than 7.5 mg of prednisone per day) within 90 days of ongoing immunosuppression.

* Patient has an untreated chronic infection or has received treatment of any uncontrolled or progressive infection with systemic antibiotics within 2 weeks prior to first CYNK-001 infusion. Prophylactic antibiotic, antiviral, and antifungal medication are permissible.
* Patient has any other organ dysfunction (CTCAE Version 5.0 Grade 3 or greater) that will interfere with the administration of the therapy according to this protocol.
* Patient has a resting left ventricular ejection fraction (LVEF) of < 40% obtained by echocardiography or multi-gated acquisition scan (MUGA).
* Patient was treated with an investigational product within 28 days of first CYNK-001 infusion. Patient must no longer be a participant in the previous interventional study at the time of CYNK-001 infusion. (Patients who are under survival follow-up or observation associated with a study are permitted, and if treatment information is collected for this period, "Investigational Study" must be used to capture the study treatment.).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2020-03-12 (Actual); Primary Completion 2023-01-20 (Actual); Study Completion 2023-04-28 (Actual)

PRIMARY OUTCOMES:
Number of Participants who experience a Dose-limiting Toxicity (DLT) in MRD positive AML patients | Day +28
  The number of participants who experience a DLT will be measured.
Number of Participants who experience a Dose-limiting Toxicity (DLT) in Relapsed/Refractory AML patients | Day +28
  The number of participants who experience a DLT will be measured.
Determine the Maximum Tolerated Dose (MTD) or Maximum Planned Dose (MPD) of CYNK-001 in MRD positive AML patients | up to 28 days
  The maximum dose safely administered for the treatment of patients with AML.
Determine the Maximum Tolerated Dose (MTD) or Maximum Planned Dose (MPD) of CYNK-001 in Relapsed/Refractory AML patients | up to 28 days
  The maximum dose safely administered for the treatment of patients with AML.
Frequency and Severity of Adverse Events (AEs) | up to 12 months
  Frequency and severity of Adverse Events will be evaluated.

SECONDARY OUTCOMES:
Number Participants who experience Minimal Residual Disease (MRD) Response | up to 12 months
  The number of participants who convert from MRD positive to MRD negative in the MRD positive arm.
Time to MRD Response | up to 12 months
  The time it takes to convert from MRD positive to MRD negative in the MRD positive arm.
Duration of MRD Response | up to 12 months
  The measure of how long participants remain MRD negative in the MRD positive arm.
Progression-free Survival (PFS) | up to 12 months
  Date of first CYNK-001 infusion to date of disease progression in the MRD positive arm.
Time to Progression (TTP) | up to 12 months
  Date of first CYNK-001 infusion to date of disease progression in the MRD positive arm.
Duration of Morphologic Complete Remission (CR) | up to 12 months
  Duration from first Morphologic CR observation to time of disease progression in the MRD positive arm.
Overall Survival (OS) | up to 12 months
  Date of first CYNK-001 infusion to date of death.
Overall Response Rate (ORR) | up to 12 months
  Defined as achievement of Complete Remission (CR), Complete Remission with incomplete (CRi) hematologic recovery, or Morphologic leukemic-free state (MLFS) in the Relapsed/Refractory AML arm.
Duration of Response (DoR) | up to 12 months
  Duration of best response in the Relapsed/Refractory AML arm.

CONTACTS AND LOCATIONS:
Overall Officials: Sharmila Koppisetti, M.D, Study Director — Celularity, Inc.
Locations (10):
- United States (10):
  - Colorado Blood Cancer Institute, Denver, Colorado
  - University of Chicago, Chicago, Illinois
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York
  - Columbia University and New York Presbyterian Hospital, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Westchester Medical Center, Valhalla, New York
  - Tennessee Oncology, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - Swedish Health Services, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dohner H, Estey E, Grimwade D, Amadori S, Appelbaum FR, Buchner T, Dombret H, Ebert BL, Fenaux P, Larson RA, Levine RL, Lo-Coco F, Naoe T, Niederwieser D, Ossenkoppele GJ, Sanz M, Sierra J, Tallman MS, Tien HF, Wei AH, Lowenberg B, Bloomfield CD. Diagnosis and management of AML in adults: 2017 ELN recommendations from an international expert panel. Blood. 2017 Jan 26;129(4):424-447. doi: 10.1182/blood-2016-08-733196. Epub 2016 Nov 28. PMID 27895058
- [Background] Levey AS, Coresh J, Greene T, Stevens LA, Zhang YL, Hendriksen S, Kusek JW, Van Lente F; Chronic Kidney Disease Epidemiology Collaboration. Using standardized serum creatinine values in the modification of diet in renal disease study equation for estimating glomerular filtration rate. Ann Intern Med. 2006 Aug 15;145(4):247-54. doi: 10.7326/0003-4819-145-4-200608150-00004. PMID 16908915